CLINICAL TRIAL: NCT00186329
Title: B-type Natriuretic Peptide for Cardio-Renal Decompensation Syndrome
Brief Title: BNP for Cardio-Renal Decompensation Syndrome (BNP-CARDS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Fowler, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SUMC79741; SPO # 29675
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Congestive Heart Failure Exacerbation; Renal Insufficiency
Keywords: Vasodilation; Congestive heart failure; Renal insufficiency; Diuresis; Serum creatinine
MeSH Terms: conditions — Renal Insufficiency; Aneurysm; Heart Failure | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: Natrecor, a recombinant form of B-type Natriuretic Peptide, made by Scios, Inc. vs. placebo

SUMMARY:
Many patients with exacerbations of heart failure have significant concomitant kidney dysfunction. The combination of these two conditions makes pharmacological management difficult. In this study, we plan to randomize patients with heart failure and kidney dysfunction to receive infusions of Natrecor (B-type Natriuretic Peptide)--which may be beneficial to the management of these two diseases--or placebo.

DETAILED DESCRIPTION:
Heart failure represents a growing epidemic in the United States. Recent figures reveal that almost 5 million people have heart failure in the U.S. alone, with an incidence (550,000 new diagnoses/year) that has increased up to threefold over the last 25 years. This growing incidence of heart failure is thought to be due to changing population demographics. Rates of major risk factors for the disease-diabetes mellitus, hypertension, and renal insufficiency--have all been steadily increasing.

Renal insufficiency causes particular difficulty for the management of heart failure. Most CHF patients have a significant degree of renal insufficiency - both because the risk factors for the two diseases are the same, but also because reduced cardiac output related to CHF leads to reduced glomerular filtration rate (GFR). Diuretics in escalating doses, a cornerstone of therapy for CHF exacerbations, can also lead to worsening renal function, a continued inability to achieve an adequate diuresis and toxicity from the agents given.

B-type Natriuretic Peptide (BNP) is a 32-amino acid peptide hormone secreted predominantly from the ventricles in response to increased pressure and volume. It has several actions in vivo, working as a diuretic, natriuretic and as a systemic pulmonary vasodilator. Natrecor is a recombinant peptide structurally identical to endogenous BNP, approved for the treatment of decompensated heart failure.

In the Vasodilation in the management of Acute Congestive Heart Failure (VMAC)trial, therapy with Natrecor resulted in improvements in pulmonary capillary wedge pressure seen within 15 minutes of starting the therapy; these improvements were significantly better than with intravenous nitroglycerine. Patients also reported a greater improvement in dyspnea with Natrecor therapy than with placebo. In a prior study, our group has demonstrated that prolonged Natrecor infusions result in improved hemodynamic parameters for Stage D heart failure patients awaiting heart transplantations.

Natrecor therapy holds theoretical value for patients with heart failure and concomitant renal insufficiency. Prior experimental work has demonstrated that BNP infusions can increase diuresis, natriuresis, and importantly, GFR in healthy subjects--all of which represent major objectives in the therapy of heart failure patients. Many have also reported the clinical experience that renal function was preserved, and diuresis/natriuresis more readily achieved in patients with heart failure exacerbations and renal insufficiency with the addition of Natrecor therapy. However, this potential use for Natrecor has not been rigorously tested.

The study is a prospective, double-blinded, placebo controlled clinical trial. Patients admitted with the medical diagnosis of CHF exacerbation and that meet study criteria will be randomized to receive Natrecor vs placebo (5% dextrose in water) intravenous infusions for 48 hrs.Randomization will occur in the pharmacy department. Patients randomized to Natrecor will receive a 2mcg/kg IV bolus, followed by a continuous infusion of 0.01mcg/kg/min. (Patients who have a net negative diuresis greater than 1 liter prior to initiation of Natrecor therapy will not receive a bolus dose given a greater risk of hypotension). Those randomized to placebo will receive a dummy bolus and infusion of the same volume of 5% dextrose in water.

100 subjects will be recruited. Inclusion criteria include inpatient admission with the diagnosis of CHF exacerbation and have a calculated creatinine clearance between 15-60 ml/min using the Cockcroft-Gault equation. Patients 18 years and older are eligible for the trial regardless of gender or ethnic background. Exclusion criteria include: hypotension (SBP< 90mmHg) at time of enrollment, severe hypertension (SBP>170 mmHg) necessitating IV vasodilator therapy, known allergy to Natrecor, history of heart transplantation, up-front use of inotropes, and contraindications to vasodilator therapy (such as severe aortic stenosis), and mental incompetence meaning inability to provide informed consent.

In addition to Stanford University Medical Center, we are beginning data collection at the VA Hospital in Palo Alto, CA.

Initial nursing management of these subjects includes every 15 minute blood pressure monitoring for hypotension. In such a case, the IV infusion will be discontinued for 36 minutes (half-life of Natrecor is 18 minutes) and then restarted. Clinical experience with Natrecor has proven this regime is usually effective.

ELIGIBILITY:
Inclusion Criteria:

* acute admission to hospital with CHF exacerbation
* calculated creatinine clearance between 15-60ml/min using the Cockroft Gault equation.

Exclusion Criteria:

* hypotension (SBP < 90mmHg)
* hypertension (SBP > 170 mmHg) necessitating vasodilator therapy
* known allergy to Natrecor
* history of heart transplantation
* contraindications to vasodilator therapy (i.e. severe aortic stenosis)
* up-front use of inotropes
* mental incompetence meaning inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-03; Study Completion 2006-10

PRIMARY OUTCOMES:
Prevention of worsened renal dysfunction (defined peak serum creatinine >20% higher than at time of admission)
Change in serum creatinine (% and absolute) from admission to discharge- or at 7 days if patient still admitted.

SECONDARY OUTCOMES:
Net negative diuresis at least 1 L/24 hours while on infusion.
Change in plasma BNP levels (meas. at admission & d/c)
Need to discontinue infusion due to symptomatic hypotension.
Total diuretic use
Resource utilization (days in hospital etc.)
Need for inotropic therapy
Readmission within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Fowler, MB, Principal Investigator — Professor, School of Medicine, Stanford University; Ronald Witteles, MD, Study Director — Cardiology Fellow, Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Background] Sackner-Bernstein JD, Skopicki HA, Aaronson KD. Risk of worsening renal function with nesiritide in patients with acutely decompensated heart failure. Circulation. 2005 Mar 29;111(12):1487-91. doi: 10.1161/01.CIR.0000159340.93220.E4. Epub 2005 Mar 21. PMID 15781736
- [Background] Sackner-Bernstein JD, Kowalski M, Fox M, Aaronson K. Short-term risk of death after treatment with nesiritide for decompensated heart failure: a pooled analysis of randomized controlled trials. JAMA. 2005 Apr 20;293(15):1900-5. doi: 10.1001/jama.293.15.1900. PMID 15840865
- [Background] Wang DJ, Dowling TC, Meadows D, Ayala T, Marshall J, Minshall S, Greenberg N, Thattassery E, Fisher ML, Rao K, Gottlieb SS. Nesiritide does not improve renal function in patients with chronic heart failure and worsening serum creatinine. Circulation. 2004 Sep 21;110(12):1620-5. doi: 10.1161/01.CIR.0000141829.04031.25. Epub 2004 Aug 30. PMID 15337695
- [Background] Colucci WS, Elkayam U, Horton DP, Abraham WT, Bourge RC, Johnson AD, Wagoner LE, Givertz MM, Liang CS, Neibaur M, Haught WH, LeJemtel TH. Intravenous nesiritide, a natriuretic peptide, in the treatment of decompensated congestive heart failure. Nesiritide Study Group. N Engl J Med. 2000 Jul 27;343(4):246-53. doi: 10.1056/NEJM200007273430403. PMID 10911006
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Witteles RM, Kao D, Christopherson D, Matsuda K, Vagelos RH, Schreiber D, Fowler MB. Impact of nesiritide on renal function in patients with acute decompensated heart failure and pre-existing renal dysfunction a randomized, double-blind, placebo-controlled clinical trial. J Am Coll Cardiol. 2007 Nov 6;50(19):1835-40. doi: 10.1016/j.jacc.2007.03.071. Epub 2007 Oct 23. PMID 17980248